CLINICAL TRIAL: NCT00386555
Title: Phase 2 Study of CP-868,596 + Docetaxel, AG-013736 + Docetaxel, or CP-868,596 + AG-013736 + Docetaxel and of Docetaxel Alone in Patients With Stage IIIb or IV Non-Small Cell Lung Cancer.
Brief Title: A Phase 2 Study in Patients With Advanced Non-Small Cell Lung Cancer Using New Agents With and Without Docetaxel.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was cancelled before patient enrollment
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5301010
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2007-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; crenolanib; Axitinib

INTERVENTIONS:
Drug: docetaxel
Drug: CP-868,596 + docetaxel
Drug: AG-013736 + docetaxel
Drug: CP-868,596 + AG-013736 + docetaxel

SUMMARY:
To determine the effectiveness of CP-868,596 + docetaxel, AG-013736 + docetaxel and CP-868,596 + AG-013736 + docetaxel in patients previously treated for non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Platinum-pretreated patients with advanced stage IIIb or IV NSCLC

Exclusion Criteria:

* Centrally-located tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Determine the anti-tumor efficacy of CP 868,596 plus docetaxel, AG 013736 plus docetaxel, CP 868,596 plus AG 013736 plus docetaxel, and docetaxel alone in patients with advanced NSCLC based on objective tumor response (CR and PR) rate

SECONDARY OUTCOMES:
Determine the safety and tolerability of the combination of daily CP 868,596 and docetaxel on an every 3 week schedule
Determine the safety and tolerability of the combination of daily AG 013736 and docetaxel on an every 3 week schedule
Determine the safety and tolerability of both CP 868,596 and AG 013736 given together with docetaxel on an every 3 week schedule
Assess additional evidence of anti-tumor activity as measured by duration of objective response, progression-free survival, and one-year survival (OS1year)
Evaluate the pharmacokinetics (PK) of AG 013736 and CP 868,596 when given together with and without docetaxel
Evaluate the PK of CP 868,596 when given in combination with docetaxel
Evaluate the PK of docetaxel when given in combination with CP 868,596, or CP 868,596 plus AG 01373

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5301010&StudyName=A+Phase+2+Study+in+Patients+with+Advanced+Non%2DSmall+Cell+Lung+Cancer+Using+New+Agents+With+and+Without+Docetaxel%2E+